CLINICAL TRIAL: NCT00654264
Title: Water Immersion in Right-Sided Heart Failure: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-29283
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Right Sided Cardiac Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Patients will have water immersion on first day and sitting in a tub without water on the second day.
  Interventions: Procedure: Water immersion
- 2 (Other): Patients will sit in a tub without water on the first day and have water immersion on the second day.
  Interventions: Procedure: Water immersion

INTERVENTIONS:
Procedure: Water immersion — Subjects will sit in tub for four hours.

SUMMARY:
This is an unblinded pilot study comparing (against a randomized control day without water immersion) the diuretic and natriuretic effects of water immersion in patients with right heart failure.

DETAILED DESCRIPTION:
Patients will be immersed in a tub for 3 hours (on one day) and neurohormones will be obtained before and after immersion. Urine will be collected for quantification and evaluation of sodium concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have right sided failure secondary to right ventricular dysfunction, pulmonary hypertension, or tricuspid regurgitation
* Age greater than 18 years of age
* Right heart catheterization within the last year to rule out left-sided failure.
* Evidence of fluid overload as indicated by 2 or more of the following: 1.) 2+ or more pitting edema of the lower extremities, 2.) scrotal or penile edema, 3.) JVP greater than or equal to 10 cm, 4.) abdominal ascites

Exclusion Criteria:

* Pulmonary capillary wedge pressure above 16 mmHg or history of elevated left ventricular filling pressures.
* Serum creatinine > 2.0
* Current use of an angiotensin I converting enzyme inhibitor or angiotensin receptor blocker will preclude participation in the RAS neurohormone portion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Diuresis | 4 hours

SECONDARY OUTCOMES:
Neurohormonal activation | 4 hours
Natriuresis | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gottlieb, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States